CLINICAL TRIAL: NCT01729650
Title: Effectiveness of a Physical Activity and Diet Program, Coordinated Between Primary Care and Mental Health, to Modify Cardiovascular Risk Factors in Patients With Schizophrenia or Bipolar Disorder (CapiCor)
Brief Title: Effectiveness of a Physical Activity and Diet Program in Patients With Psychotic Disorder (CapiCor)
Acronym: CapiCor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Carlos III Health Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PI11/01861
Record Dates: First submitted 2012-11-14; First posted 2012-11-20 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-08

CONDITIONS: Schizophrenic Disorders; Schizoaffective Disorders; Bipolar Disorders
Keywords: Psychotic Disorders,; Heart Diseases
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Bipolar Disorder; Heart Diseases | interventions — Restraint, Physical

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physical and diet educational group (Experimental): group educational PA program (basically walking) of 24 sessions over 12 weeks, and diet (16 sessions in the first 8 weeks), carried out by mental health nurses.
  Interventions: Behavioral: Physical and diet educational group
- Usual clinical care (No Intervention)

INTERVENTIONS:
Behavioral: Physical and diet educational group — educational group of: physical activity program (basically walking) of 24 sessions over 12 weeks, and diet (16 sessions in the first 8 weeks, carried out by mental health nurses.
  Arms: Physical and diet educational group

SUMMARY:
The aim is to evaluate the effectiveness of an intervention based on a program of physical activity and diet coordinated between primary care teams (PCT) and Mental Health Centres (MHC) to modify the weekly physical activity (PA) amount, body mass index (BMI) and waist circumference in patients with severe mental disorder diagnoses. To assess changes in cardiovascular risk, quality of life and lifestyles, secondarily. Methods: A randomized clinical trial with a control group, of one year of follow-up, carried out in four MHC Barcelona and Santa Coloma, and PCT of reference. The investigators studied patients aged 18 - 65 years old, diagnosed with schizophrenia, schizoaffective or bipolar disorder, with antipsychotic medication and a low level of PA. 240 patients will be selected in each group (difference to be detected in the BMI:> 1.89 kg/m2; common SD: 6.2, 30% loss). Intervention: group educational PA program (basically walking) of 24 sessions over 12 weeks, and diet (8 sessions in the first 8 weeks) by nurses and specialists in PA. Key measurements: level of PA (IPAQ questionnaire), physical examinations: BMI, waist circumference, blood pressure, cardiovascular risk, quality of life (SF-36), smoking habits, dietary habits (PREDIMED questionnaire), analytical parameters: cholesterol , triglycerides, blood glucose. Evaluations will be masked and conducted at 0, 3, 6 and 12 months. Analysis of variance for repeated measures to adjust for differences attributable to the effect of the intervention for potential confounders: pharmacological treatment, care level of intervention and mental state.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 65 years old,
* understand Catalan or Spanish
* will be located for at least twelve months.
* Psychiatric disorders with ICD-10 diagnosis codes: F20*, F31* and F25*.
* Taking an antipsychotic drug at, a least, three months
* Low physical activity level

Exclusion Criteria:

* Active addiction to psychoactive drugs, except tobacco.
* Pregnancy
* Diseases that doesn't allow physical activity
* Psychotic acute exacerbation in the last month

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Actual)
Dates: Start 2012-06; Primary Completion 2015-03 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in weekly level of physical activity (IPAQ questionnaire), | : the outcome measure is studied at 3, 6 and 12 months
Body mass index (kg/m²) | : the outcome measure is studied at 3, 6 and 12 months
waist circumference (cm) | : the outcome measure is studied at 3, 6 and 12 months

SECONDARY OUTCOMES:
blood pressure (mm hg) | the outcome measure is studied at 3, 6 and 12 months
cardiovascular risk with the Regicor coronary risk to 10 years | the outcome measure is studied at 3, 6 and 12 months
Quality of life (SF-36 questionnaire) | the outcome measure is studied at 3, 6 and 12 months
Smoking habits: smoker/ ex-smoker/no-smoker. Number of cigarettes per day. | the outcome measure is studied at 3, 6 and 12 months
Dietary habits (PREDIMED questionnaire) | the outcome measure is studied at 3, 6 and 12 months
Analytical parameters: cholesterol , triglycerides, blood glucose mg/100 ml. | the outcome measure is studied at 3, 6 and 12 months

OTHER OUTCOMES:
Clinical Global Impression, CGI | the outcome measure is studied at 3, 6 and 12 months
BPRS (Brief Psychiatric Rating Scale) | the outcome measure is studied at 3, 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: MARIA-ISABEL FERNANDEZ-SAN-MARTIN, PH, Principal Investigator — Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina
Locations (1):
- Jordi Gol i Gurina Foundation, Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Masa-Font R, Fernandez-San-Martin MI, Martin Lopez LM, Alba Munoz AM, Oller Canet S, Martin Royo J, San Emeterio Echevarria L, Olona Tabuena N, Ibarra Jato M, Barroso Garcia A, Gonzalez Tejon S, Tajada Vitales C, Diaz Mujica B, Vinas Cabrera L, Sanchis Catalan R, Salvador Barbarroja T. The effectiveness of a program of physical activity and diet to modify cardiovascular risk factors in patients with severe mental illness after 3-month follow-up: CAPiCOR randomized clinical trial. Eur Psychiatry. 2015 Nov;30(8):1028-36. doi: 10.1016/j.eurpsy.2015.09.006. Epub 2015 Oct 30. PMID 26521223